CLINICAL TRIAL: NCT02289482
Title: A Double-Blind, Randomized, Placebo-Controlled, Continuation Single Dose Escalation Study to Investigate the Safety, Tolerability and Pharmacokinetics of GSK2838232 With and Without Ritonavir, and to Evaluate Different Formulations of GSK2838232, in Healthy Subjects
Brief Title: A Single Dose Pharmacokinetic (PK) and Safety Study of GSK2838232 With and Without Ritonavir (RTV) Conducted in Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study prematurely terminated due to safety concerns leading to clinical hold
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200912
Record Dates: First submitted 2014-11-10; First posted 2014-11-13 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: Ritonavir; Safety; Continuation Single Dose Escalation; GSK2838232
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — Ritonavir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK2838232 Part A: Single Dose Escalation (Experimental): During Part A, subjects will receive GSK2838232/ placebo (3:1) in 4-period (period 1: GSK2838232 200mg, period 2: GSK2838232 500mg), single dose escalation design. Subjects randomized to placebo will receive placebo in all four periods. Following completion of Period 2 PK assessments at 96hr post-dose, subjects will begin daily dosing of RTV 100mg (period 3: GSK2838232 20 mg + RTV 100 mg, period 4: GSK2838232 50 mg + RTV 100 mg) for a total of 26 days.
  Interventions: Drug: GSK2838232 PIB (SDD); Drug: Placebo; Drug: Ritonavir
- GSK2838232 Part B: Single Dose, 3-Period Crossover, Relative B (Experimental): During Part B, subjects will receive GSK2838232/ placebo, in an open-label, unbalanced, 3-period, cross-over design; subjects will be randomized (1:1) to each sequence. The relative bioavailability of single 100 mg doses of powder in a bottle (PIB) Active Pharmaceutical Ingredient (API) of GSK2838232 versus PIB Spray-Dried Dispersion (SDD) will be assessed (Period 1: SDD GSK2838232 100 mg vs GSK2838232 API 100 mg; period 2: GSK2838232 API 100 mg Vs SDD GSK2838232 100 mg ). A single dose of GSK2838232 will be co-administered on the 10th day of RTV dosing (period 3:GSK2838232 10 mg + RTV 100 mg); RTV dosing will continue for an additional 4 days (total of 14 days).
  Interventions: Drug: GSK2838232 PIB (SDD); Drug: GSK2838232 PIB (API); Drug: Placebo; Drug: Ritonavir

INTERVENTIONS:
Drug: GSK2838232 PIB (SDD) — GSK2838232 will be available as oral suspension dispersion in hydromellulose acetate succinate bulk powder/10, 20, 50, 200 and 500 mg in part A, while 100 mg in Part B. GSK2838232 will be administered orally once daily (QD) as single doses in the morning following an overnight fast of at least 10 hours.
Drug: GSK2838232 PIB (API) — GSK2838232 will be available as oral suspension bulk powder/100 mg in Part B. GSK2838232 will be administered orally QD as single doses in the Morning following an overnight fast of at least 10 hours.
  Arms: GSK2838232 Part B: Single Dose, 3-Period Crossover, Relative B
Drug: Placebo — Matching placebo of Suspension to active dose, administered orally QD as single doses in the morning following an overnight fast of at least 10 hours.
Drug: Ritonavir — Ritonavir will be available as white film-coated ovaloid tablets of 100 mg tablet/100mg. Ritonavir will be administered orally, once daily in Part A, Period 3 Days 1-14 and Period 4 from Days 1-12 and will be administer orally once daily in Part B for 9 days prior to dosing in Period 3 and on Days 10-14 of Period 3.

SUMMARY:
This study investigates the safety, tolerability and PKs of GSK2838232 with and without Ritonavir, and to evaluate different formulations of GSK2838232 in healthy subjects. This study will evaluate higher single and RTV boosted doses to support continued clinical development of GSK2838232 at clinically relevant doses, and subsequently in those infected with HIV in a dose ranging phase 2 study. The study is conducted in 2 parts: Part A and Part B, study Part A and Part B may be conducted in parallel. Approximately 20 healthy subjects will be enrolled into the study, 8 in Part A and 12 in Part B. Part A is a double-blind, randomized, placebo-controlled, 4-period, single dose escalation design. Subjects will be randomized 3:1 to receive GSK2838232 or placebo. Subjects randomized to placebo will receive placebo in all four periods. Following completion of Period 2 PK assessments at 96hr post-dose, subjects will begin daily dosing of RTV 100mg for a total of 26 days.

Part B is a randomized, open-label, unbalanced, 3-period, cross-over design; subjects will be randomized 1:1 to each sequence. The relative bioavailability of single 100mg doses of powder in a bottle (PIB) active pharmaceutical ingredient (API) of GSK2838232 versus PIB spray-dried dispersion (SDD) will be assessed. A single dose of GSK2838232 will co-administered on the 10th day of RTV dosing; RTV dosing will continue for an additional 4 days (total of 14 days). Subjects will have a screening visit within 30 days prior to first dose and a follow-up visit 7-14 days after the last dose.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 55 years of age inclusive, at the time of signing the informed consent
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator in consultation with the Medical Monitor if required agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* A Creatinine clearance (CLcr) >80 millilitre per minute (mL/min) as determined by Cockcroft-Gault equation where age is in years, weight (Wt) is in kg, and serum creatinine (Scr) is in units of milligram / decilitre (mg/dL); CLcr (mL/min) = (140 - age) * Wt / (72 * Scr) (times 0.85 if female).
* Body weight >= 50 kilogram (kg [110 pounds {lbs}]) for men and >= 45 kg (99 lbs) for women and body mass index (BMI) within the range 18.5-31.0 kilogram per meter square kg/m^2 (inclusive)
* Male or Female; Female subject of non-reproductive potential : is eligible to participate if she is not pregnant (as confirmed by a negative serum or urine human chorionic gonadotrophin (hCG) test), not lactating, and at least one of the following conditions applies: Pre-menopausal females with one of the following: Documented tubal ligation, Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, Hysterectomy, Documented Bilateral Oophorectomy; Postmenopausal defined as 12 months of spontaneous amenorrhea in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause (refer to laboratory reference ranges for confirmatory levels). Females on hormone replacement therapy (HRT) must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. Male subjects with female partners of child bearing potential must comply with the following contraception requirements from the time of first dose of study medication until one week after the last dose of study medication. a) Vasectomy with documentation of azoospermia, b) Male condom plus partner use of one of the contraceptive options below: Contraceptive subdermal implant that meets the standard operating procedure (SOP) effectiveness criteria including a <1% rate of failure per year, as stated in the product label, Intrauterine device or intrauterine system that meets the SOP effectiveness criteria including a <1% rate of failure per year, as stated in the product label, Oral Contraceptive, either combined or progestogen alone Injectable progestogen, Contraceptive vaginal ring, Percutaneous contraceptive patches. These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.

Exclusion Criteria:

* Alanine aminotransferase and bilirubin >1.5xupper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Subjects who have asthma or a history of asthma.
* Medical history of cardiac arrhythmias or cardiac disease or a family and personal history of long QT syndrome.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* Regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* Screening or baseline cardiac troponin I greater than the 99% cutoff (>.045 nanogram/ milliliter [ng/mL] by the Dimension Vista Cardiac troponin assay).
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 56 days.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Exclusion Criteria for 24-Hour Screening Holter: Any symptomatic arrhythmia (except isolated extra systoles), Sustained cardiac arrhythmias (such as atrial fibrillation or flutter, supraventricular tachycardia (>=10 consecutive beats), complete heart block). Non-sustained or sustained ventricular tachycardia (defined as >= 3 consecutive ventricular ectopic beats). Any conduction abnormality (including but not specific to left or right incomplete or complete bundle branch block, atrioventricular (AV) block [2nd degree or higher], Wolff-Parkinson-White [WPW] syndrome etc.). Sinus Pauses > 3 seconds. 300 or more supraventricular ectopic beats in 24 hours. 250 or more ventricular ectopic beats in 24 hours.
* Any clinically significant abnormal echocardiogram finding. Abnormal echocardiogram findings should be discussed with the Medical Monitor prior to enrolment.
* Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination): Heart rate <45 and >100 beats per minute (bpm) (Males); <50 and >100 bpm (females); For both Males and Females: PR Interval <120 and >220 msec, QRS duration <70 and >120 millisecond (msec); QTc interval (Fridericia's) >450 msec. Notes: A heart rate from 100 to 110 bpm can be rechecked by ECG or vitals within 30 minutes to verify eligibility. Evidence of previous myocardial infarction (Does not include ST segment changes associated with repolarization). Any conduction abnormality (including but not specific to left or right complete bundle branch block, AV block [2nd degree or higher], WPW syndrome). Sinus Pauses > 3 seconds. Any significant arrhythmia which, in the opinion of the principal investigator or GlaxoSmithKline medical monitor, will interfere with the safety for the individual subject. Non-sustained or sustained ventricular tachycardia (>= 3 consecutive ventricular ectopic beats).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-11-17 (Actual); Primary Completion 2015-03-10 (Actual); Study Completion 2015-03-10 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) assessments | Up to approximately 7 weeks
  Safety was assessed by monitoring AE and serious AEs (SAE). AEs and SAEs will be collected from the start of Study Treatment until the follow-up contact
Safety assessed by laboratory evaluations | Up to approximately 7 weeks
  Laboratory evaluations will include hematology, clinical chemistry, urinalysis assessments
Vital signs assessments | Up to approximately 7 weeks
  Vital signs will be measured in semi-supine position after 10 minutes rest and will include systolic and diastolic blood pressure and pulse rate.
Electrocardiogram (ECG) parameters assessments | Up to approximately 7 weeks
  Triplicate or Single 12-lead ECGs will be obtained at each timepoint during the study after a 10 minute rest using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTc intervals.
Composite PK profile of GSK2838232, , with and without RTV for Part A and Part B | During Part A: Day 1 to Day 5 (Period 1 & 2), Day 10-Day 15 (Period 3), Day 8 - Day 13 (Period 4). During Part B: Day 1 to Day 4 (Period 1 & 2), Day 10-Day 14 (Period 3)
  PK assessments will include: area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC 0-infinity), area under the concentration-time curve over the dosing interval (AUC 0-t), concentration at 24 hours post dose (C24), oral clearance (CL/F), maximum observed concentration (Cmax), last quantifiable concentration (Clast), time of occurrence of Cmax (tmax), time of last observed concentration (tlast), terminal phase half-life (t1/2), and time of first quantifiable concentration (tlag).
Composite PK profile of GSK2838232 to assess the relative bioavailability of the PIB API suspension versus PIB SDD suspension (Part B) | During Part B: Day 1 to Day 4 (Period 1 & 2), Day 10-Day 14 (Period 3)
  PK assessments will include: GSK2838232 AUC(0-infinity), Cmax
Composite PK profile of GSK2838232 to assess single dose proportionality of GSK2838232 with and without steady-state RTV (Part A) | During Part A: Day 1 to Day 5 (Period 1 & 2), Day 10-Day 15 (Period 3), Day 8 - Day 13 (Period 4).
  PK assessments will include: GSK2838232 AUC(0 - infinity), AUC(0-t) and Cmax

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

REFERENCES:
- See also: Results for study 200912 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/200912?search=study&search_terms=200912#rs